CLINICAL TRIAL: NCT01875120
Title: Prospective Observational Study to Evaluate Somatic Symptom Load and Anxiety Sensitivity as Risk Factors for Postoperative Nausea and Vomiting (PONV)
Brief Title: Study to Evaluate Anxiety Sensitivity and Somatic Symptoms as Risk Factors for PONV
Acronym: somPONV
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Rita Laufenberg-Feldmann, M.D., Deputy senior physician, head of clinical trial unit, Johannes Gutenberg University Mainz
Other Study IDs: 837.327.12 (8428-F)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Anxiety; Somatoform Disorders
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Anxiety Disorders; Somatoform Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Female patients with increased risk to experience PONV.

SUMMARY:
This prospective observational study aims to evaluate the influence of somatic symptom load and anxiety sensitivity as risk factors for the occurrence of postoperative nausea and vomiting (PONV). Physiological and psychological variables are assessed in female patients with an increased risk for PONV prior to a planned surgical intervention with a 33-item questionnaire composed of the ASI-3 and the PHQ-15. Postoperative evaluation includes the occurrence of nausea and vomiting in the first 24 hours after surgery. It is hypothesized that patients with high sum scores for somatic symptom load (measured with the Patient Health Questionnaire, PHQ-15) and with increased levels for anxiety sensitivity (measured with the Anxiety Sensitivity Index, ASI-3) experience more frequently postoperative nausea and vomiting (PONV) than patients with low scores in both self-rating instruments.

ELIGIBILITY:
Inclusion Criteria:

* female patients 18-75 years
* non-smokers
* must be able to give written informed consent
* planned surgical intervention requiring hospitalisation
* not included in another clinical trial

Exclusion Criteria:

* emergency intervention
* total intravenous anesthesia (TIVA) with propofol
* disability to give written informed consent
* physical or psychic disorders requiring permanent psycho-social care
* no German language skills

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients in a universitary hospital who are scheduled for elective surgery in general anesthesia (planned interventions in general surgery, orthopedia, traumatology, gynecology, neurosurgery (except intracranial interventions)and who present with an increased risk to experience postoperative nausea and vomiting.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of postoperative nausea and vomiting (PONV). | PONV is assessed in the first 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Gutenberg University Medical Center, Department of Anesthesiology, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Apfel CC, Roewer N, Korttila K. How to study postoperative nausea and vomiting. Acta Anaesthesiol Scand. 2002 Sep;46(8):921-8. doi: 10.1034/j.1399-6576.2002.460801.x. PMID 12190791
- [Background] Asmundson GJ, Taylor S. Role of anxiety sensitivity in pain-related fear and avoidance. J Behav Med. 1996 Dec;19(6):577-86. doi: 10.1007/BF01904905. PMID 8970916
- [Background] Barsky AJ, Wyshak G, Klerman GL. The somatosensory amplification scale and its relationship to hypochondriasis. J Psychiatr Res. 1990;24(4):323-34. doi: 10.1016/0022-3956(90)90004-a. PMID 2090830
- [Background] Kisely S, Goldberg D, Simon G. A comparison between somatic symptoms with and without clear organic cause: results of an international study. Psychol Med. 1997 Sep;27(5):1011-9. doi: 10.1017/s0033291797005485. PMID 9300507
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Lee YY, Kim KH, Yom YH. Predictive models for post-operative nausea and vomiting in patients using patient-controlled analgesia. J Int Med Res. 2007 Jul-Aug;35(4):497-507. doi: 10.1177/147323000703500409. PMID 17697527
- [Background] Van den Bosch JE, Moons KG, Bonsel GJ, Kalkman CJ. Does measurement of preoperative anxiety have added value for predicting postoperative nausea and vomiting? Anesth Analg. 2005 May;100(5):1525-1532. doi: 10.1213/01.ANE.0000149325.20542.D4. PMID 15845719
- [Background] Watcha MF, White PF. Postoperative nausea and vomiting. Its etiology, treatment, and prevention. Anesthesiology. 1992 Jul;77(1):162-84. doi: 10.1097/00000542-199207000-00023. PMID 1609990
- [Derived] Laufenberg-Feldmann R, Muller M, Ferner M, Engelhard K, Kappis B. Is 'anxiety sensitivity' predictive of postoperative nausea and vomiting?: A prospective observational study. Eur J Anaesthesiol. 2019 May;36(5):369-374. doi: 10.1097/EJA.0000000000000979. PMID 30865002